CLINICAL TRIAL: NCT01564862
Title: A Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, Active-Referenced, Flexible Dose Study on the Efficacy of Lu AA21004 on Cognitive Dysfunction in Adult Subjects With Major Depressive Disorder (MDD)
Brief Title: Efficacy of Lu AA21004 on Cognitive Dysfunction in Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LuAA21004_202; 2011-005298-22 (EudraCT Number); U1111-1126-0091 (Registry Identifier: WHO)
Record Dates: First submitted 2012-03-26; First posted 2012-03-28 (Estimated); Results first posted 2015-02-05 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Depressive Disorder, Major
Keywords: Drug Therapy
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Vortioxetine; Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vortioxetine (Lu AA21004) QD (Experimental): Vortioxetine (Lu AA21004) 10 mg, capsules, orally, once daily for one week; then dose adjustment to a maximum 20 mg, capsules, orally, once daily for up to 7 weeks.
  Interventions: Drug: vortioxetine (Lu AA21004)
- Duloxetine QD (Active Comparator): Duloxetine 60 mg, capsules, orally, for up to 8 weeks. Duloxetine 30 mg, capsule, orally, once daily for 1 week taper-down period.
  Interventions: Drug: Duloxetine
- Placebo QD (Placebo Comparator): Placebo matching capsules, orally, once daily for up to 9 weeks (includes 1 week taper down period).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: vortioxetine (Lu AA21004) — Lu AA21004 capsules
  Arms: Vortioxetine (Lu AA21004) QD
Drug: Duloxetine — Duloxetine capsules
  Other Names: Cymbalta
  Arms: Duloxetine QD
Drug: Placebo — Placebo matching capsules
  Arms: Placebo QD

SUMMARY:
The purpose of this study is to evaluate the effects of Lu AA21004, once daily (QD), on cognitive dysfunction in patients with major depressive disorder.

DETAILED DESCRIPTION:
Lu AA21004 is under codevelopment by Takeda Global Research & Development Center, Inc. and H. Lundbeck A/S for the treatment of MDD.

This study will consist of a screening period within 10 days of the Baseline Visit followed by an 8-week double-blind treatment period and a one-week taper down period.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. The participant has recurrent MDD as the primary diagnosis according to Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria (classification code 296.3x). The current MDE should be confirmed using the Mini International Neuropsychiatric Interview (MINI) V6.0.0.
4. The participant has received prescribed treatment for a previous episode of depression.
5. The participant has a MADRS total score ≥26 at both the screening and baseline visits.
6. Participant reports subjective cognitive dysfunction (such as difficulty concentrating, slow thinking, and difficulty in learning new things or remembering things).
7. The reported duration of the current major depressive episode (MDE) is at least 3 months
8. The participant is a man or woman between 18 and 65 years old, inclusive.
9. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to routinely use adequate contraception from signing of the informed consent throughout the duration of the study and for 30 days after completion of the study.

Exclusion Criteria:

1. The participant has previously participated in this study.
2. The participant has a history of severe drug allergy or hypersensitivity, or known hypersensitivity to any of the excipients of the investigational medicinal product (IMP).
3. The participant has known hypersensitivity to duloxetine.
4. The participant has hereditary problems of fructose intolerance, glucose-galactose malabsorption, or sucrose-isomaltase insufficiency.
5. The participant is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in the conduct of this study (e.g., spouse, parent, child, sibling) or may consent under duress.
6. The participant has a score ≥70 on the DSST (numbers correct) at the Baseline Visit.
7. The participant is, in the opinion of the investigator, not able to complete the neuropsychological tests validly at the Baseline Visit.
8. If female, the participant is pregnant or lactating or intending to become pregnant before, during, or within 30 days after participating in this study; or intending to donate ova during such time period.
9. The participant has 1 or more of the following:

   1. Any current psychiatric disorder other than MDD as defined in the DSM-IV-TR (as assessed by the MINI Version 6.0.0).
   2. Current or history of attention deficit hyperactivity disorder (ADHD), pervasive developmental disorder, manic or hypomanic episode, schizophrenia, or any other psychotic disorder, including major depression with psychotic features, mental retardation, organic mental disorders, or mental disorders due to a general medical condition as defined in the DSM-IV-TR.
   3. Current diagnosis of alcohol or other substance abuse or dependence (excluding nicotine or caffeine) as defined in the DSM-IV-TR that has not been in sustained full remission for at least 2 years prior to Screening. (Participant must also have negative urine drug screen prior to Baseline).
   4. Presence or history of a clinically significant neurological disorder (including epilepsy).
   5. Neurodegenerative disorder (Alzheimer's disease, Parkinson's disease, multiple sclerosis, Huntington's disease, etc).
   6. Any DSM-IV Axis II disorder that might compromise the study.
10. The participant has any other disorder for which the treatment takes priority over treatment of MDD or is likely to interfere with study treatment or impair treatment compliance.
11. The participant has physical, cognitive, or language impairment of such severity as to adversely affect the validity of the data derived from the neuropsychological tests.
12. The participant is diagnosed with reading disability (dyslexia).
13. The participant has a significant risk of suicide according to the investigator's clinical judgment or has a score ≥5 on item 10 (suicidal thoughts) of the MADRS or has made a suicide attempt in the previous 6 months.
14. The participant, in the opinion of the investigator, poses a risk of harm to others.
15. The participant has initiated formal cognitive or behavioral therapy, systemic psychotherapy within less than 6 months of study screening, or has plans to initiate such therapy during the study.
16. The participant has received electroconvulsive therapy, vagal nerve stimulation, or repetitive transcranial magnetic stimulation within 6 months prior to Screening.
17. The current depressive symptoms are considered by the investigator to have been resistant to 2 adequate antidepressant treatments of at least 6 weeks duration each at the recommended dose.
18. The participant has a history of moderate or severe head trauma (for example, loss of consciousness for more than 1 hour) or other neurological disorders or systemic medical diseases that are, in the opinion of the investigator, likely to affect central nervous system functioning.
19. The participant has a previous history of cancer that had been in remission for less than 5 years prior to the first dose of investigational drug. This criterion does not include those participants with basal cell or stage I squamous cell carcinoma of the skin.
20. The participant has a clinically significant unstable illness, for example, hepatic impairment or renal insufficiency, or cardiovascular, pulmonary, gastrointestinal, endocrine, neurological, rheumatologic, immunologic, infectious, skin and subcutaneous tissue disorders, or metabolic disturbance.

    Note: For the purposes of this protocol, the following conditions are considered unstable due to the potential impact on assessment of MDD response and/or cognitive status: pain disorders, chronic fatigue syndrome, fibromyalgia, obstructive sleep apnea, and known cases of HIV, HBV, and HCV
21. The participant has a known history of or currently has increased intraocular pressure or is at risk of acute narrow-angle glaucoma.
22. The participant is required to take excluded medications or it is anticipated that the participant will require treatment with at least 1 of the disallowed concomitant medications during the study evaluation period as specified in the Excluded Medications Section.
23. The participant has received any investigational compound <30 days before Screening or 5 half-lives prior to Screening.
24. The participant has clinically significant abnormal vital signs as determined by the investigator.
25. The subject has thyroid stimulating hormone (TSH) outside the normal range at the Screening Visit.

    Note: If TSH value is outside the normal range, a free T4 will be obtained. Subjects who have elevated TSH but normal T4 (i.e. subclinical hypothyroidism) will be excluded. For subjects who are on thyroid hormone replacement therapy, a lower TSH with normal T4, are eligible to participate in the study only if there are no clinical symptoms of hypothyroidism .
26. The participant has 1 or more laboratory value outside the normal range, based on the blood or urine samples taken at the Screening Visit, that are considered by the investigator to be clinically significant; or the participant has any of the following values at the Screening Visit:

    1. A serum creatinine value >1.5 times the upper limits of normal (×ULN).
    2. A total serum total bilirubin value >1.5×ULN.
    3. A serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) value >2×ULN.
27. The participant has an abnormal electrocardiogram (ECG) as determined by the central reader and confirmed as clinically significant by the investigator.
28. The participant has a disease or takes medication that, in the opinion of the investigator, could interfere with the assessments of safety, tolerability, or efficacy.
29. The participant, in the opinion of the investigator, is unlikely to comply with the clinical study protocol or is unsuitable for any reason.
30. The participant has been previously exposed to LuAA21004 compound.
31. The participant has a history of lack of response to previous adequate treatment with duloxetine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 602 (Actual)
Dates: Start 2012-04; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director Clinical Science, Study Director — Takeda
Locations (92):
- United States (62):
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Bellflower, California
  - Carson, California
  - Cerritos, California
  - Glendale, California
  - Imperial, California
  - Los Angeles, California
  - Norwalk, California
  - Oakland, California
  - Paramount, California
  - San Bernardino, California
  - Santa Ana, California
  - Wildomar, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Norwalk, Connecticut
  - Lauderhill, Florida
  - Miami, Florida
  - Orlando, Florida
  - Sanford, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Chicago, Illinois
  - Hoffman Estates, Illinois
  - Naperville, Illinois
  - Oak Brook, Illinois
  - Skokie, Illinois
  - Indianapolis, Indiana
  - Prairie Village, Kansas
  - Shreveport, Louisiana
  - Baltimore, Maryland
  - Haverhill, Massachusetts
  - St Louis, Missouri
  - North Platte, Nebraska
  - Las Vegas, Nevada
  - Buffalo, New York
  - New York, New York
  - Staten Island, New York
  - Avon Lake, Ohio
  - Beachwood, Ohio
  - Garfield Heights, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Allentown, Pennsylvania
  - Norristown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Columbia, South Carolina
  - Franklin, Tennessee
  - Memphis, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - The Woodlands, Texas
  - Orem, Utah
  - Salt Lake City, Utah
  - Kirkland, Washington
  - Seattle, Washington
  - Brown Deer, Wisconsin
  - Milwaukee, Wisconsin
- Bulgaria (6):
  - Kazanlak
  - Novi Iskar
  - Pleven
  - Plovdiv
  - Sofia
  - Tzerova Koria
- Finland (3):
  - Helsinki
  - Kuopio
  - Turku
- Germany (8):
  - Berlin
  - Bochum
  - Chemnitz
  - Hanover
  - München
  - Schwerin
  - Westerstede
  - Wiesbaden
- Poland (4):
  - Bialystok
  - Leszno
  - Lodz
  - Torun
- Russia (5):
  - Nizhny Novgorod
  - Saint Petersburg
  - Smolensk
  - Stavropol
  - Yekaterinburg
- Ukraine (4):
  - Kharkiv
  - Kyiv
  - Luhansk
  - Ternopil

REFERENCES:
- [Derived] Jacobson W, Zhong W, Nomikos GG, Christensen MC, Kurre Olsen C, Harvey PD. Effects of vortioxetine on functional capacity across different levels of functional impairment in patients with major depressive disorder: a University of California, San Diego Performance-based Skills Assessment (UPSA) analysis. Curr Med Res Opin. 2020 Jan;36(1):117-124. doi: 10.1080/03007995.2019.1657692. Epub 2019 Aug 29. PMID 31422713
- [Derived] Christensen MC, Sluth LB, McIntyre RS. Validation of the University of California San Diego Performance-based Skills Assessment (UPSA) in major depressive disorder: Replication and extension of initial findings. J Affect Disord. 2019 Feb 15;245:508-516. doi: 10.1016/j.jad.2018.11.034. Epub 2018 Nov 5. PMID 30439678
- [Derived] Christensen MC, Loft H, McIntyre RS. Vortioxetine improves symptomatic and functional outcomes in major depressive disorder: A novel dual outcome measure in depressive disorders. J Affect Disord. 2018 Feb;227:787-794. doi: 10.1016/j.jad.2017.11.081. Epub 2017 Nov 16. PMID 29689693
- [Derived] Keefe RSE, Nomikos G, Zhong W, Christensen MC, Jacobson W. A Subgroup Analysis of the Impact of Vortioxetine on Functional Capacity, as Measured by UPSA, in Patients with Major Depressive Disorder and Subjective Cognitive Dysfunction. Int J Neuropsychopharmacol. 2018 May 1;21(5):442-447. doi: 10.1093/ijnp/pyy020. PMID 29546401
- [Derived] Christensen MC, Munro V. Cost per successfully treated patient for vortioxetine versus duloxetine in adults with major depressive disorder: an analysis of the complete symptoms of depression and functional outcome. Curr Med Res Opin. 2018 Apr;34(4):593-600. doi: 10.1080/03007995.2017.1416952. Epub 2018 Jan 16. PMID 29235884
- [Derived] Harvey PD, Jacobson W, Zhong W, Nomikos GG, Cronquist Christensen M, Kurre Olsen C, Merikle E. Determination of a clinically important difference and definition of a responder threshold for the UCSD performance-based skills assessment (UPSA) in patients with major depressive disorder. J Affect Disord. 2017 Apr 15;213:105-111. doi: 10.1016/j.jad.2017.02.014. Epub 2017 Feb 14. PMID 28213121

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 80 investigative sites in Bulgaria, Finland, Germany, Poland, Russia Federation, Ukraine.and the United States from 09 April 2012 to 05 February 2014
Pre-assignment Details: Participants with a diagnosis of major depressive disorder were enrolled equally in 1 of 3 treatment groups, once a day placebo, 10 to 20 mg flexible dose of vortioxetine, or 60 mg duloxetine.
Groups:
- Vortioxetine (Lu AA21004): Vortioxetine (Lu AA21004) 10 mg, capsules, orally, once daily for one week; then dose adjustment to a maximum 20 mg, capsules, orally, once daily for up to 7 weeks.
- Duloxetine: Duloxetine 60 mg, capsules, orally, for up to 8 weeks. Duloxetine 30 mg, capsule, orally, once daily for 1 week taper-down period.
- Placebo: Placebo matching capsules, orally, once daily for up to 9 weeks (includes 1 week taper down period).
Period: Overall Study
Arm/Group | Vortioxetine (Lu AA21004) | Duloxetine | Placebo
Started | 198 | 210 | 194
Received Treatment | 196 | 207 | 191
Completed | 168 | 176 | 164
Not Completed | 30 | 34 | 30
Not completed — Pretreatment Event or Adverse Event | 6 | 12 | 6
Not completed — Major Protocol Deviation | 3 | 3 | 4
Not completed — Lost to Follow-up | 10 | 8 | 6
Not completed — Voluntary Withdrawal | 9 | 6 | 8
Not completed — Lack of Efficacy | 1 | 5 | 6
Not completed — Other reason(s) | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vortioxetine (Lu AA21004) | Duloxetine | Placebo | Total
Number analyzed (Participants) | 198 | 210 | 194 | 602
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (12.21) | 45.7 (11.46) | 45.0 (12.07) | 45.0 (11.90)
Age, Customized [Number; unit: participants]
  ≤ 55 years | 158 | 164 | 152 | 474
  > 55 years | 40 | 46 | 42 | 128
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135 | 138 | 119 | 392
  Male | 63 | 72 | 75 | 210
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 8 | 7 | 15 | 30
  Non-Hispanic and Non- Latino | 90 | 104 | 82 | 276
  Not-Specified | 100 | 99 | 97 | 296
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian (or White, including Hispanic) | 169 | 176 | 171 | 516
  Black | 28 | 27 | 20 | 75
  Asian | 1 | 6 | 1 | 8
  American Indian or Alaska Native | 0 | 1 | 2 | 3
Height [Mean (Standard Deviation); unit: cm] | 168.2 (9.17) | 169.7 (9.14) | 169.0 (9.43) | 169.0 (9.25)
Weight [Mean (Standard Deviation); unit: kg] | 81.84 (22.068) | 81.68 (20.965) | 80.96 (20.316) | 81.50 (21.099)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.86 (7.334) | 28.39 (7.312) | 28.27 (6.354) | 28.51 (7.018)
Smoking Classification [Number; unit: participants]
  Never Smoked | 95 | 109 | 105 | 309
  Current Smoker | 73 | 68 | 56 | 197
  Past Smoker | 30 | 33 | 33 | 96
Alcohol Consumption [Number; unit: participants]
  Never | 89 | 84 | 87 | 260
  Once Monthly or Less Often | 67 | 73 | 51 | 191
  Once a Week | 23 | 31 | 29 | 83
  2 to 6 Times per Week | 15 | 19 | 24 | 58
  Daily | 4 | 3 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 8 in the Digit Symbol Substitution Test (DSST)
Description: The DSST assesses relative contributions of speed, memory, executive function and visual scanning. Participants are required to copy symbols that are paired with simple geometric shapes or numbers within a specific time for a total possible score of 0 to 133. Higher scores-correct number of symbols reflects greater objective cognitive functioning. An increase in score represents an improvement in an integrated measure of cognitive function. An Analysis of Covariance (ANCOVA) model was used with treatment and center as fixed factors and the Baseline value as a covariate.
Time Frame: Baseline and Week 8
Population: Full Analysis Set included all randomized participants who received at least one dose of study drug and had at least 1 valid post-baseline value for assessment of primary efficacy. Participants with scores of > 70 at Baseline were excluded.
Measure: Least Squares Mean (Standard Error); unit: Correct symbols
Arm/Group | Vortioxetine (Lu AA21004) | Duloxetine | Placebo
Number analyzed (Participants) | 175 | 187 | 167
Correct symbols | 4.60 (0.530) | 4.06 (0.511) | 2.85 (0.542)
Statistical Analysis 1: Comparison: Vortioxetine (Lu AA21004) vs Placebo; Test type: Superiority or Other; p = 0.019, ANCOVA — P-value was from an ANCOVA model with treatment and center as fixed factors and the baseline value as a covariate; LS mean difference = 1.75, 95% CI 2-sided [0.28 to 3.21], Standard Error of Mean 0.744
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.099, ANCOVA — P-value was from an ANCOVA model with treatment and center as fixed factors and the baseline value as a covariate; LS mean difference = 1.21, 95% CI 2-sided [-0.23 to 2.65], Standard Error of Mean 0.733
Statistical Analysis 3: Comparison: Vortioxetine (Lu AA21004) vs Duloxetine; Test type: Superiority or Other; p = 0.460, ANCOVA — P-value was from an ANCOVA model with treatment and center as fixed factors and the baseline value as a covariate; LS mean difference = 0.54, 95% CI 2-sided [-0.89 to 1.96], Standard Error of Mean 0.725

2. Secondary Outcome: Change From Baseline to Week 8 in the Perceived Deficits Questionnaire (PDQ) Attention/Concentration and Planning/Organization Subscore
Description: PDQ is a patient-rated scale designed to subjectively assess cognitive dysfunction, comprising four 5-item subscales: Attention/Concentration, Retrospective Memory, Prospective Memory, and Planning/Organization for a total possible score of 0 to 40. The subscale Attention/Concentration is the sum of items 1, 5, 9, 13, and 17 with a range of 0-20; while the subscale Planning/Organization is the sum of items 4, 8, 12, 16, and 20 with the score range of 0 to 20. The scores of the subscales Attention/Concentration and Planning/Organization were summed. Higher scores reflect greater participant-perceived cognitive dysfunction in the domains identified. A decrease in score represents an improvement in subjective cognitive function in the domains identified. A Mixed Model Repeated Measures (MMRM) model was used with baseline*week, center, week, treatment and week*treatment as factors in the analysis.
Time Frame: Baseline and Week 8
Population: Participants from the Full Analysis Set, all randomized participants who received at least one dose of study drug and had at least 1 valid post-baseline value for assessment of primary efficacy,with data available for analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Vortioxetine (Lu AA21004) | Duloxetine | Placebo
Number analyzed (Participants) | 169 | 179 | 160
score on a scale | -8.9 (0.55) | -9.3 (0.53) | -6.3 (0.57)
Statistical Analysis 1: Comparison: Vortioxetine (Lu AA21004) vs Placebo; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis — P-value was from a MMRM model with baseline*week, center, week, treatment and week*treatment as factors in the analysis; LS Mean difference = -2.6, 95% CI 2-sided [-4.1 to -1.0], Standard Error of Mean 0.78
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value was from a MMRM model with baseline*week, center, week, treatment and week*treatment as factors in the analysis; LS mean difference = -3.0, 95% CI 2-sided [-4.5 to -1.5], Standard Error of Mean 0.77

3. Secondary Outcome: Clinical Global Impressions-Improvement (CGI-I) Score at Week 8
Description: The CGI-I assesses the clinician's impression of the subject's state of mental illness improvement and consists of one question for the investigator: "Compared to his condition at the start of the study, how much has this patient changed?" which is rated on a seven-point scale (1=very much improved; 2=much improved; 3=minimally improved; 4=no change relative to baseline; 5=minimally worse; 6= much worse; 7=very much worse). Higher scores indicate greater worsening of illness. Values closest to 1 for this outcome measure indicate the greatest improvement of symptoms. A MMRM model was used with baseline*week, center, week, treatment and week*treatment as factors in the analysis.
Time Frame: Baseline, Week 8
Population: Participants from the Full Analysis Set, all randomized participants who received at least one dose of study drug and had at least 1 valid post-baseline value for assessment of primary efficacy, with data available for analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Vortioxetine (Lu AA21004) | Duloxetine | Placebo
Number analyzed (Participants) | 169 | 179 | 161
score on a scale | 2.349 (0.0852) | 2.235 (0.0826) | 2.639 (0.0872)
Statistical Analysis 1: Comparison: Vortioxetine (Lu AA21004) vs Placebo; Test type: Superiority or Other; p = 0.017, Mixed Models Analysis — P-value was from a MMRM model with baseline*week, center, week, treatment and week*treatment as factors in the analysis; LS Mean difference = -0.290, 95% CI 2-sided [-0.528 to -0.052], Standard Error of Mean 0.1211
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value was from a MMRM model with baseline*week, center, week, treatment and week*treatment as factors in the analysis; LS mean difference = -0.404, 95% CI 2-sided [-0.638 to -0.169], Standard Error of Mean 0.1194

4. Secondary Outcome: Change From Baseline to Week 8 in the Trail Making Test (TMT-A)
Description: The TMT is a two-part cognitive test. TMT-A assesses cognitive processing speed and consists of 25 circles distributed over a sheet of paper. Participants have 4 minutes to connect the circles as quickly as possible, without lifting the pen or pencil from the paper. Tester informs participant immediately whenever they make an error and allows for corrections by participants. Lower scores represent better speed of processing. A decrease in score over the study represents an improvement in speed in processing. An ANCOVA model was used with treatment and center as fixed factors and the baseline value as a covariate.
Time Frame: Baseline and Week 8
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | Vortioxetine (Lu AA21004) | Duloxetine | Placebo
Number analyzed (Participants) | 173 | 180 | 162
seconds | -7.70 (0.980) | -8.06 (0.955) | -6.65 (1.009)

5. Secondary Outcome: Change From Baseline to Week 8 in the Trail Making Test B (TMT-B)
Description: The TMT is a two-part cognitive test. TMT-B assesses executive functioning and consists of 25 circles distributed over a sheet of paper. Participants have 4 minutes to connect the circles as quickly as possible, without lifting the pen or pencil from the paper. Tester informs participant immediately whenever they make an error and allows for corrections by participants. Lower score for TMT-B represents better executive function. A decrease in score over the study represents an improvement in executive function. An ANCOVA model was used with treatment and center as fixed factors and the Baseline value as a covariate.
Time Frame: Baseline and Week 8
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | Vortioxetine (Lu AA21004) | Duloxetine | Placebo
Number analyzed (Participants) | 157 | 170 | 157
seconds | -18.73 (2.096) | -14.60 (2.011) | -9.06 (2.101)

6. Secondary Outcome: Change in Time From Baseline to Week 8 in the Stroop Test
Description: The STROOP test assesses the ability to inhibit a prepotent response to reading words while performing a task that requires attention control. It comprises of 2 sheets with 50 words each, up to 50 correct responses for each of the congruent and incongruent Stroop tests. Participants have 4 minutes to name the ink color of each word. Lower time to complete the test indicates better performance. Higher number of correct responses indicates better responses. A decrease in the time to complete the tests and an increase in the number of correct responses both indicate improvement over the course of the study. An ANCOVA model was used with treatment and center as fixed factors and the Baseline value as a covariate.
Time Frame: Baseline and Week 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Vortioxetine (Lu AA21004) | Duloxetine | Placebo
Number analyzed (Participants) | 175 | 187 | 167
seconds
  Congruent (n=174,187,167) | -3.30 (1.086) | -4.54 (1.044) | -4.37 (1.105)
  Incongruent (n=172,186,166) | -8.17 (1.560) | -9.83 (1.498) | -8.11 (1.586)

7. Secondary Outcome: Change From Baseline to Week 8 in the Groton Maze Learning Test (GMLT)
Description: The GMLT measures executive functioning and spatial problem solving. Participants learn a hidden pathway through a maze of 10 x 10 grid of tiles on a computer touch screen using step-by-step guess, with trial and error feedback after each step. Once the pathway is learned, participants repeat the same pathway four more times. It usually takes 5-6 minutes to administer this test. Lower score equals better performance. A decrease in score over the course of the study indicates improved executive function.
  An ANCOVA model was used with treatment and center as fixed factors and the Baseline value as a covariate.
Time Frame: Baseline and Week 8
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Errors
Arm/Group | Vortioxetine (Lu AA21004) | Duloxetine | Placebo
Number analyzed (Participants) | 169 | 179 | 159
Errors | -5.43 (1.355) | -5.16 (1.314) | -3.49 (1.397)

8. Secondary Outcome: Change From Baseline to Week 8 in the Detection Task (DT)
Description: The DT is a computerized test that measures simple reaction time and psychomotor speed. The task requires participants to respond by pressing a "yes" button as soon as an onscreen playing card is turned over and is red, and by pressing a "no" button if the card is not red. It takes 2 minutes to be administered. There is no minimum or maximum scores since it is a time-based assessment. Lower score equals better performance. A decrease in score over the course of the study indicates improved speed of processing and psychomotor function. An ANCOVA model was used with treatment and center as fixed factors and the Baseline value as a covariate.
Time Frame: Baseline and Week 8
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Log10 milliseconds
Arm/Group | Vortioxetine (Lu AA21004) | Duloxetine | Placebo
Number analyzed (Participants) | 175 | 182 | 167
Log10 milliseconds | -0.050 (0.0080) | -0.039 (0.0078) | -0.033 (0.0082)

9. Secondary Outcome: Change From Baseline to Week 8 in the Identification Task (IT)
Description: The IT measured choice reaction time: the participant pressed a "yes" button whenever an onscreen playing card turned face up and was red, or a "no" button if the card was not red. The IT took on average 2 minutes to complete. Lower scores equal better performance. A decrease in score over the course of the study indicates improved visual attention/vigilance. An ANCOVA model was used with treatment and center as fixed factors and the Baseline value as a covariate.
Time Frame: Baseline and Week 8
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Log10 milliseconds
Arm/Group | Vortioxetine (Lu AA21004) | Duloxetine | Placebo
Number analyzed (Participants) | 175 | 182 | 167
Log10 milliseconds | -0.037 (0.0060) | -0.030 (0.0059) | -0.024 (0.0062)

10. Secondary Outcome: Change From Baseline to Week 8 in the One-Back Task
Description: The One-Back test measures the cognitive domain of attention and working memory through yes or no responses to 30 trials. The task requires participants to report when a stimulus item presented serially is the same as an item one step back from the item at hand for a total correct responses 0 to 100. It usually takes 2-3 minutes to be administered. Higher scores equal better performance. An increase in score over the course of the study indicates improved attention/working memory. An ANCOVA model was used with treatment and center as fixed factors and the Baseline value as a covariate.
Time Frame: Baseline and Week 8
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Log 10 milliseconds
Arm/Group | Vortioxetine (Lu AA21004) | Duloxetine | Placebo
Number analyzed (Participants) | 175 | 182 | 167
Log 10 milliseconds | -0.028 (0.0062) | -0.024 (0.0060) | -0.022 (0.0063)

11. Secondary Outcome: Proportion of Cognitive Dysfunction Improvement Due to Improvement of Depression
Description: Improvement of Cognitive Dysfunction is determined using the change from Baseline to Week 8 in the Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score and the Digital Symbol Substitution Test (DSST) total number of correct symbols. The MADRS is a 10-item clinician rated scale to measure overall severity of depressive symptoms (such as apparent sadness, reported sadness, inner tension) rated on a 7-point Likert scale from 0 (symptoms absent) to 6 (severe depression). The DSST assesses relative contributions of speed, memory, executive function and visual scanning. The proportion of direct effect from treatment = DSST difference / (DSST difference + coefficient*MADRS difference).
Time Frame: Baseline and Week 8
Population: Full Analysis Set included all participants who were randomized, received at least 1 dose of study drug, and had at least 1 valid post-baseline value for assessment.
Measure: Number; unit: proportion of direct effect
Arm/Group | Vortioxetine (Lu AA21004) | Duloxetine
Number analyzed (Participants) | 175 | 187
proportion of direct effect | 75.66 | 48.69

12. Secondary Outcome: Change From Baseline to Week 8 in the MADRS Total Score
Description: MADRS is a 10-item clinician rated scale to measure overall severity of depressive symptoms (such as apparent sadness, reported sadness, inner tension) rated on a 7-point Likert scale from 0 (symptoms absent) to 6 (severe depression) with a total possible score range from 0 to 60. Higher scores indicate greater severity of symptoms. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Week 1, Week 4 and Week 8
Population: Full Analysis Set included all randomized participants who received at least one dose of study drug and had at least 1 valid post-baseline value for assessment of primary efficacy. Last Observation Carried Forward.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vortioxetine (Lu AA21004) | Duloxetine | Placebo
Number analyzed (Participants) | 175 | 187 | 167
score on a scale
  Change at Week 1 | -3.7 (4.80) | -4.6 (5.29) | -3.4 (5.03)
  Change at Week 4 | -9.8 (6.85) | -11.6 (7.94) | -8.0 (7.98)
  Change at Week 8 | -14.3 (8.97) | -15.5 (9.23) | -12.3 (9.64)

13. Secondary Outcome: Percentage of Participants With MADRS Response at Week 8
Description: MADRS is a 10-item clinician rated scale to measure overall severity of depressive symptoms (such as apparent sadness, reported sadness, inner tension) rated on a 7-point Likert scale from 0 (symptoms absent) to 6 (severe depression) with a total possible score range from 0 to 60. Higher scores indicate greater severity of symptoms. MADRS Response was defined as a ≥50% decrease in MADRS Total Score from Baseline.
Time Frame: Baseline and Week 8
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | Vortioxetine (Lu AA21004) | Duloxetine | Placebo
Number analyzed (Participants) | 175 | 187 | 167
percentage of participants | 50.9 | 54.5 | 41.3

14. Secondary Outcome: Percentage of Participants in MADRS Remission at Week 8
Description: MADRS is a 10-item clinician rated scale to measure overall severity of depressive symptoms (such as apparent sadness, reported sadness, inner tension) rated on a 7-point Likert scale from 0 (symptoms absent) to 6 (severe depression) with a total possible score range from 0 to 60. Higher scores indicate greater severity of symptoms. MADRS Remission was defined as a MADRS total score ≤10.
Time Frame: Week 8
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | Vortioxetine (Lu AA21004) | Duloxetine | Placebo
Number analyzed (Participants) | 175 | 187 | 167
percentage of participants | 30.3 | 33.7 | 21.6

15. Secondary Outcome: Change From Baseline to Week 8 in the Clinical Global Impressions-Severity (CGI-S) Score
Description: The CGI-S assesses the clinician's impression of the subject's current state of mental illness and consists of one question for the investigator: "Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?" which is rated on a seven-point scale (1=normal, not ill at all; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill). A MMRM model with baseline*week, center, week, treatment and week*treatment as factors was used for analyses.
Time Frame: Baseline, Week 1, Week 4 and Week 8
Population: Participants from the Full Analysis Set, all randomized participants who received at least one dose of study drug and had at least 1 valid post-baseline value for assessment of primary efficacy,with data available for analysis. Repeated Measures Analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Vortioxetine (Lu AA21004) | Duloxetine | Placebo
Number analyzed (Participants) | 175 | 187 | 167
score on a scale
  Change from Baseline at Week 1 (n=174, 187,167) | -0.289 (0.0426) | -0.353 (0.0410) | -0.243 (0.0435)
  Change from Baseline at Week 4 (n=173,184,165) | -0.951 (0.0678) | -1.170 (0.0656) | -0.617 (0.0693)
  Change from Baseline at Week 8 (n=169,179,161) | -1.546 (0.0886) | -1.698 (0.0859) | -1.225 (0.0906)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug and no more than 30 days after the last dose of study drug (Up to 12 Weeks)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Vortioxetine (Lu AA21004) | Duloxetine | Placebo
Serious Adverse Events (participants affected / at risk) | 1/196 | 1/207 | 2/191
Other Adverse Events (participants affected / at risk) | 73/196 | 84/207 | 41/191
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vortioxetine (Lu AA21004) (N=196) | Duloxetine (N=207) | Placebo (N=191)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vortioxetine (Lu AA21004) (N=196) | Duloxetine (N=207) | Placebo (N=191)
Nausea (Gastrointestinal disorders) | 40 | 43 | 8
Diarrhoea (Gastrointestinal disorders) | 11 | 6 | 5
Dry mouth (Gastrointestinal disorders) | 6 | 16 | 9
Nasopharyngitis (Infections and infestations) | 7 | 8 | 11
Decreased appetite (Metabolism and nutrition disorders) | 3 | 12 | 1
Headache (Nervous system disorders) | 20 | 24 | 16
Dizziness (Nervous system disorders) | 6 | 11 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.